CLINICAL TRIAL: NCT07053982
Title: 18F]-FES PET in the Detection and Characterization of Endometriosis Lesions
Brief Title: Use of a New Diagnostic Tool in the Detection and Characterization of Endometriosis Lesions
Acronym: ENDO-TEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/23/0622; 2025-520637-24-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-10; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Endometriosis
Keywords: Endometriosis; Estrogen receptors; Pain; [18F]-FES PET/CT
MeSH Terms: conditions — Endometriosis; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endometriosis Patients Undergoing Surgery for Severe Pain Management (EVA ≥ 4) (Experimental)
  Interventions: Procedure: Preoperative [18F]-FES PET/CT Imaging and Estrogen Receptor Expression Analysis in Endometriosis Surgery
- Endometriosis Patients Undergoing Surgery for Infertility Without Severe Pain (EVA < 4) (Experimental)
  Interventions: Procedure: Preoperative [18F]-FES PET/CT Imaging and Estrogen Receptor Expression Analysis in Endometriosis Surgery

INTERVENTIONS:
Procedure: Preoperative [18F]-FES PET/CT Imaging and Estrogen Receptor Expression Analysis in Endometriosis Surgery — This study includes preoperative [18F]-FES PET/CT imaging to assess estrogen receptor expression in endometriosis patients undergoing laparoscopic or robot-assisted surgery. Pain levels will be evaluated using VAS, BPI, HADS, and SF-36 scales. Immunohistochemistry and quantitative mRNA expression analysis (ESR1, ESR2, GPER) will be performed on excised lesions using Tissue Microarray. This approach aims to correlate PET/CT imaging findings with histological and molecular data, distinguishing it from standard surgical interventions.

SUMMARY:
Diagnostic wandering is one of the characteristics of endometriosis due to great anatomical and clinical variability but also due to poorly relevant diagnostic examinations. [18F]-FES PET/CT could on the one hand improve diagnosis by showing greater sensitivity than MRI and on the other hand make it possible to quantify and characterize the expression of ER from diagnosis and thus helping to guide therapeutic care. We will thus attempt to correlate the intensity of [18F]-FES PET/CT with the expression of estrogen receptors and the intensity of pain.

DETAILED DESCRIPTION:
Endometriosis is a chronic estrogen-dependent gynecological condition that leads to impaired overall quality of life due to infertility and associated pain. Diagnostic wandering is one of the characteristics of endometriosis due to great anatomical and clinical variability but also due to poorly relevant diagnostic examinations. There are several anatomo-clinical pathological entities. Thus, its painful symptoms vary greatly in its location and intensity. MRI, the reference examination for diagnosis but operator dependent, shows imperfect sensitivity. The diagnosis and characterization of lesions must therefore be improved. We know that 17β-estradiol, a key hormone for lesion growth, can also be produced locally by endometriotic tissue. The hypothesis according to which this local accumulation of estrogens plays an important role in the development of lesions by modulating the expression of RE must be studied. The use of new tools to study estrogen receptor expression should be evaluated at diagnosis. A new examination, [18F]-FES PET/CT, could on the one hand improve diagnosis by showing greater sensitivity than MRI and on the other hand make it possible to quantify and characterize the expression of the ER from the diagnosis and thus help to guide therapeutic care. [18F]-FES PET/CT is a non-invasive, operator-independent method that visualizes and quantifies ER expression in multiple tumors. Some studies have shown that [18F]-FES uptake correlates well with ER expression measured by immunohistochemistry staining. We will thus attempt to correlate the intensity of [18F]-FES PET/CT with the expression of estrogen receptors and the intensity of pain.

ELIGIBILITY:
Inclusion Criteria:

Cases:

- Painful patients with a VAS ≥ 4 treated surgically for painful symptoms related to endometriosis;

Controls:

* Patient with a VAS < 4 treated surgically for endometriosis in the context of infertility;
* Age > 18 years;
* Patient who provided informed consent;
* Patients who underwent a preoperative MRI and were not contraindicated for [18F]-FES PET/CT;
* Patient who underwent surgery mid-cycle;
* Affiliation to a social security scheme

Exclusion Criteria:

* Patient treated for endometriosis without surgery;
* Pregnant patient
* Patient taking hormone therapy
* Menopausal patient
* Hypersensitivity to the active substance (Fluoroestradiol (18F)) or to any of the excipients
* Patient under legal protection
* Claustrophobic patient

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Quantification of Estrogen Receptor Overexpression in Endometriotic Lesions Using SUV on [18F]-FES PET/CT | Preoperative assessment at mid-cycle, before surgery and without concurrent hormonal treatment.
  Estrogen receptor (ER) overexpression in endometriotic lesions will be assessed using the Standardized Uptake Value (SUV) on preoperative [18F]-FES PET/CT imaging. Each lesion's SUV will be quantified and compared within patients and between groups with high pain levels (VAS ≥ 4) and low or no pain (VAS < 4). ER overexpression is defined as increased [18F]-FES uptake compared to background levels. The correlation between SUV values and pain severity will be analyzed to determine whether ER overexpression is associated with symptomatic burden. Higher SUV values indicate greater ER expression.

SECONDARY OUTCOMES:
Characterization of Lesion Staining by Immunohistochemistry and In Situ Hybridization: Intensity and Receptor Expression by Anatomical Location. | From tissue collection at surgery to completion of immunohistochemical and in situ hybridization analyses (approximately 4 weeks post-surgery).
  Lesions were analyzed using immunohistochemistry (IHC) and in situ hybridization to characterize receptor expression patterns (ERα, ERβ, GPER) and staining intensity. Tissue microarrays (TMA) from 20 patients were used to standardize analysis. IHC staining was performed with specific antibodies against ERα (SP1) and ERβ (CWK-F12 (DSHB)), while in situ hybridization was conducted using Bio-Techne probes targeting ESR1, ESR2, and GPER mRNA. Staining intensity and receptor expression were assessed for each lesion and compared across anatomical locations. Correlation with [18F]-FES PET/CT imaging and clinical symptomatology was also evaluated.
Sensitivity of [18F]-FES PET/CT Compared to MRI for Diagnosing Superficial and Deep Endometriotic Lesions by Anatomical Location. | From completion of MRI and [18F]-FES PET/CT imaging (performed within 4 weeks prior to surgery) to histopathological analysis of lesions obtained during surgery (within 4 weeks post-imaging); total assessment period: up to 8 weeks per participant
  The sensitivity of [18F]-FES PET/CT in detecting superficial and deep endometriotic lesions will be compared to that of MRI. Lesions will be classified based on their anatomical location. Sensitivity will be calculated as the proportion of true positive lesions detected by each imaging modality, using surgical and histopathological findings as the reference standard. The diagnostic performance of PET/CT and MRI will be analyzed for different lesion types and locations to assess their respective accuracy in detecting endometriosis.
Association Between [18F]-FES SUV Intensity, Estrogen Receptor Expression (IHC), and Pain Severity (VAS Score) | From the date of [18F]-FES PET/CT imaging (≤4 weeks before surgery) to the date of surgery and completion of pain assessments (VAS and BPI) and histopathological analysis of surgical samples; total duration of assessment per participant : up to 8 weeks
  The association between [18F]-FES standardized uptake value (SUV) intensity, estrogen receptor (ER) expression assessed by immunohistochemistry (IHC), and pain severity will be analyzed. ER expression will be evaluated using specific antibodies for ERα and ERβ, and quantified based on staining intensity. Pain severity will be assessed using the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst possible pain). Correlations will be determined to assess the relationship between tracer uptake, receptor expression, and pain perception
Correlation Between Estrogen Receptor Expression in IHC/ISH and Pain Intensity (VAS) in Endometriosis | From surgery (biopsy collection) to completion of pain assessment and histological analysis; up to 8 weeks.
  Estrogen receptor expression (ERα, ERβ, GPER) will be assessed in endometriotic lesions using immunohistochemistry (IHC) and in situ hybridization (ISH). Staining intensity will be scored semi-quantitatively (e.g., 0 to 3). Pain severity will be measured using the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst possible pain). A correlation analysis will be conducted to evaluate the relationship between receptor expression scores and VAS scores. The unit of measure will be the correlation coefficient between IHC/ISH scores and VAS units (0-10 scale).
Correlation Between Estrogen Receptor mRNA Expression and Pain Intensity (VAS) in Endometriosis | From surgery (biopsy collection) to completion of ISH and VAS assessments; up to 8 weeks.
  Estrogen receptor mRNA expression (ESR1, ESR2, GPER) will be quantified in endometriotic lesions using in situ hybridization (ISH). Expression levels will be evaluated based on signal intensity scores derived from probe hybridization. Pain severity will be measured using the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst pain). A statistical correlation will be assessed between the mRNA expression signal intensity scores and VAS values. The unit of measure will be the correlation coefficient quantifying the relationship between receptor expression levels and reported pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Ariane WEYL, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Toulouse, Rangueil Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No